CLINICAL TRIAL: NCT06983509
Title: Registry of Pre-mixed Solutions in Critically Ill Patients on the Continuous Renal Replacement Therapy (PrioR): a Multicenter, Prospective Real-world
Brief Title: Registry of Pre-mixed Solutions in Critically Ill Patients on the Continuous Renal Replacement Therapy
Acronym: PrioR
Status: Recruiting | Type: Observational
Sponsor: Vantive Health LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: BXU605703
Record Dates: First submitted 2025-04-23; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Renal Insufficiency
Keywords: Continuous renal replacement therapy; Hemofiltration replacement solutions
MeSH Terms: conditions — Renal Insufficiency | interventions — Phosphorus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CRRT with Regiocit/Prismasol 2/Biphozyl: Critically ill adult patients receiving CRRT with at least one of the three pre-mixed solutions (Regiocit, Prismasol 2, or Biphozyl).
  The mode of therapy, solute formulations, flow rates, fluid removal rate, and length of therapy is selected by the physician responsible for managing treatment, depending on the clinical condition of the patient, as well as the patient's fluid, electrolyte, acid-base, and glucose balance. An initial CRRT dose of 30 mL/kg/h is advised to achieve the recommended effluent volume of 20 to 25 mL/kg/h. Patients weighing more than 100 kg may not exceed a CRRT dose of 4 L/h.
  Interventions: Drug: Regiocit; Drug: Biphozyl; Drug: Prismasol 2

INTERVENTIONS:
Drug: Regiocit — Regiocit can be used as a replacement fluid for CRRT with RCA. It will be used in pre-dilution mode only.
  At least 200 mL of post-replacement solution is recommended to minimize clotting in the de-aeration chamber. A replacement/dialysate solution with 22 to 26 mEq/L bicarbonate buffer is advised as the first choice. A higher concentration of bicarbonate may be required in severe cases of acidosis. The use of a non-calcium-containing dialysate or replacement fluid is advised. The rate of administration depends on the targeted citrate dose and the prescribed flow rate. The pre-filter infusion rate of Regiocit will be indexed to the blood flow rate (BFR) to achieve a target blood citrate concentration of 3 to 4 mmol/L. A BFR between 100 to 180 mL/min will be advised; a lower BFR can minimize patient citrate exposure, particularly in patients with lower body weight.
  Other Names: Sodium citrate replacement solution
Drug: Biphozyl — Biphozyl is used as a replacement fluid during CRRT. It is injected into the extracorporeal circuit before (pre-dilution) or after (post-dilution) the filter. After the initiation of RRT, Biphozyl is used for late treatment of the acute condition when pH, potassium, and phosphate concentrations return to normal. Biphozyl can also be used if any other buffer is in use or during RCA.
  The volume and rate of administration of Biphozyl depend on the blood concentration of phosphate and other electrolytes, acid-base balance, body fluid balance, and overall clinical condition of the patient. The volume of replacement fluid given also depends on the expected intensity (dosage) of treatment.
  Other Names: Phosphorus/sodium bicarbonate replacement solution
Drug: Prismasol 2 — Prismasol 2 is used as a replacement fluid during CRRT. It is injected into the extracorporeal circuit before (pre-dilution) or after (post-dilution) the filter.
  The volume and rate of administration of Prismasol 2 depend on the blood concentration of electrolytes, acid-base balance, fluid balance, and overall clinical condition of the patient. The volume of replacement fluid administered also depends on the required intensity (dosage) of the treatment.
  Other Names: Sodium bicarbonate replacement solution

SUMMARY:
This is a multicenter, prospective, registry study. By collecting relevant demographic information and clinical data of patients receiving continuous renal replacement therapy (CRRT) with pre-mixed solutions, the clinical applicability of pre-mixed solutions will be evaluated in critically ill patients in real-world clinical settings.

This study will be carried out in approximately 10 study sites in China. Patient data will be collected to evaluate the clinical applicability of pre-mixed solutions.

DETAILED DESCRIPTION:
Treatment observation period: From initiation of the first CRRT with sponsored pre-mixed solutions to cessation of the pre-mixed solutions. The duration of this period can be up to 10 days.

Follow-up period: from the cessation of sponsored pre-mixed solutions to Day 30 after starting treatment with the pre-mix solutions.

ELIGIBILITY:
Inclusion Criteria:

* 18 ≤ age < 80 years old.
* Patients admitted to the intensive care unit (ICU) and in need of CRRT.
* Patients are willing to receive CRRT with at least one of three pre-mixed solutions:

Regiocit, Biphozyl, or Prismasol 2.

Exclusion Criteria:

* Patients with chronic kidney failure who are receiving maintenance dialysis.
* Patients expected to require the premixed solution for less than 24 hours.
* Patients who are allergic or have contraindications to components of pre-mixed solutions, as determined by the investigators.
* Patients who have participated in other interventional studies within the last 30 days.
* Patients who are pregnant, breastfeeding, or abortus imminence.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill adult patients who require CRRT with one of the following pre-mixed solutions: Regiocit, Biphozyl, or Prismasol 2.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Filter Lifespan - Duration | From initiation of 1st CRRT with sponsored solutions until mandatory replacement at 72 hours, death, access problems, filter or circuit clotting, filter membrane rupture, elective stopping of the filter, or achievement of treatment goals, whichever first
  The duration of filter use during the use of pre-mixed solutions
Filter Lifespan - Replacement or Discontinuation | From initiation of 1st CRRT with sponsored solutions until mandatory replacement at 72 hours, death, access problems, filter or circuit clotting, filter membrane rupture, elective stopping of the filter, or achievement of treatment goals, whichever first
  The reasons for replacing or discontinuing the filter during the use of pre-mixed solutions
Electrolyte and Acid-Base Indicators - Calcium | Within 4 hours before the start of CRRT (baseline), 2h ± 1h, 6h ± 2h after the start of CRRT, and daily after 24h of CRRT initiation until the end of use of the pre-mixed solutions during the 1st CRRT session.
  Serum ionized calcium, total calcium and post-filter ionized calcium
Electrolyte and Acid-Base Indicators - Potassium | Within 4 hours before the start of CRRT (baseline), and daily after 24h of CRRT initiation until the end of use of the pre-mixed solutions during the 1st CRRT session.
  Potassium
Electrolyte and Acid-Base Indicators - Sodium | Within 4 hours before the start of CRRT (baseline), and daily after 24h of CRRT initiation until the end of use of the pre-mixed solutions during the 1st CRRT session.
  Sodium
Electrolyte and Acid-Base Indicators - Phosphate | Within 4 hours before the start of CRRT (baseline), and daily after 24h of CRRT initiation until the end of use of the pre-mixed solutions during the 1st CRRT session.
  Phosphate
Electrolyte and Acid-Base Indicators - Magnesium | Within 4 hours before the start of CRRT (baseline), and daily after 24h of CRRT initiation until the end of use of the pre-mixed solutions during the 1st CRRT session.
  Magnesium
Electrolyte and Acid-Base Indicators - Bicarbonate | Within 4 hours before the start of CRRT (baseline), and daily after 24h of CRRT initiation until the end of use of the pre-mixed solutions during the 1st CRRT session.
  Bicarbonate
Electrolyte and Acid-Base Indicators - pH | Within 4 hours before the start of CRRT (baseline), and daily after 24h of CRRT initiation until the end of use of the pre-mixed solutions during the 1st CRRT session.
  Blood pH value
User experience of the pre-mixed solutions | At the end of the study, i.e., Day 30 post treatment
  A questionnaire about the preparation time, ease of operation, and additional workload when using the pre-mixed solutions will be provided to the investigators to collect information on user experience.
Severe bleeding events | From initiation of the 1st CRRT with sponsored solutions until Day 7 post treatment
  1. The requirement to transfuse 400 mL of whole blood or more than 2U of red blood cell suspension/concentrated red blood cells due to bleeding in a single time.
  2. Bleeding that requires reoperation
  3. New-onset intracranial hemorrhage without traumatic events.
Citrate accumulation | From initiation of the 1st CRRT with sponsored solutions until Day 7 post treatment
  Defined as a total/ionized calcium ratio in serum >2.5, with metabolic acidosis (as determined by the investigator)

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - Beijing Chao-yang Hospital, Capital Medical University, Beijing
  - Beijing Anzhen Hospital, Capital Medical University, Beijing
  - Xuanwu Hospital Capital Medical University, Beijing
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing
  - The First People's Hospital of Guangzhou, Guangzhou
  - Zhujiang Hospital, Southern Medical University, Guangzhou
  - Zhejiang Provincial People's Hospital, Hangzhou
  - ZhongShan Hospital Fudan University, Shanghai
  - Shanghai East Hospital, Shanghai
  - Zhongnan Hospital, Wuhan University, Wuhan

IPD SHARING:
Plan to Share IPD: Undecided